CLINICAL TRIAL: NCT03816436
Title: The Impact of Clavicular Length Restoration in the Treatment of Non-unions of Clavicular Midshaft and Lateral Fractures
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00120; ch19Mueller
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Clavicular Length
Keywords: clavicle non-unions; plate treatment of clavicular fractures; cortical bone grafting of clavicular fractures; clavicular midshaft non- union; clavicular lateral non- union; clavicular shortening
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Follow- up (FU) assessment on clavicular non- union: clavicular midshaft and lateral non- union treated by plate and iliac crest bone grafting
  Interventions: Other: Follow- up (FU) assessment

INTERVENTIONS:
Other: Follow- up (FU) assessment — Follow- up (FU) assessment (clinical examination and patient questionnaires) at least 24 months after surgery (clavicular midshaft and lateral non- union treated by plate and iliac crest bone grafting)

SUMMARY:
Evaluating the impact of plate treatment and cortical bone grafting of clavicular midshaft and lateral non- unions on restoration of clavicular length and bony healing and its association with functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* clavicular midshaft and lateral non- union treated by plate and iliac crest bone grafting
* minimal follow- up of two years after surgery
* written informed consent

Exclusion Criteria:

* legal incompetence
* non- union of pathologic fractures
* current pregnancy
* German language barrier to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients surgically treated at the Schulthess Clinic (KWS) and at the University Hospital Basel (USB) for internal fixation with a plate and using iliac bone graft of clavicular non- unions.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Clavicula shortening (cm) | one assessment at least 24 months after clavicular surgery by plate and iliac crest bone grafting
  Clavicula shortening (cm) based on Imaging assessment (x-ray, ultrasound), dichotomous outcome with shortening less or equal 2 cm (yes/no).

SECONDARY OUTCOMES:
Constant Murley score (CS) | one assessment at least 24 months after clavicular surgery by plate and iliac crest bone grafting
  tool for assessment of shoulder function: Range of Motion (ROM) of shoulder (degree), abduction strength (kg), Quality of Life (QoL) questionnaire. The different scales are summed and normalized to 0=worst to 100=best.
Subjective shoulder pain (NRS) | one assessment at least 24 months after clavicular surgery by plate and iliac crest bone grafting
  Patient rates pain at rest and at motion of the treated shoulder on numeric scale ranging from 0 (no pain) to 10 (maximum possible pain)
Subjective shoulder value (SSV) | one assessment at least 24 months after clavicular surgery by plate and iliac crest bone grafting
  based on a single question answered subjectively by Patient: "What is the overall percent value of your shoulder if a completely normal shoulder represents 100%?"
Simple shoulder test (SST) | one assessment at least 24 months after clavicular surgery by plate and iliac crest bone grafting
  12 items questionnaire to assess restrictions in activities of daily living (ADL) related to impaired shoulder function; response in dichotomous manner (yes/no)
Quality of Life (QoL) | one assessment at least 24 months after clavicular surgery by plate and iliac crest bone grafting
  assessed by Quality of Life EuroQoL 5D-5L Instrument (EQ-5D-5L); the descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Mueller, PD Dr. med, Principal Investigator — Orthopädische Universitätsklinik Basel
Locations (2):
- Switzerland (2):
  - Department of Orthopaedics, Basel
  - Schulthess Klinik Zürich, Zurich